CLINICAL TRIAL: NCT06156007
Title: Effect of Progressive Muscle Relaxation Exercise on RLS Severity, Quality of Life and Sleep Quality in Menopausal Women with Restless Legs Syndrome (RLS): a Randomized Controlled Study
Brief Title: Effect of Progressive Muscle Relaxation Exercises in Menopausal Women Experiencing RLS.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Pinar Akbas, assistant professor doctor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: menopause
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Restless Legs Syndrome
Keywords: restless legs syndrome; menopause; progressive muscle relaxation exercises
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Intervention Model Description: The research was planned as a single-center, parallel randomized controlled experimental study with stratified randomization (mild-moderate, severe-very severe) and pretest-posttest control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- progressive muscle relaxation exercises (Experimental): Women will be given one-time progressive muscle relaxation exercise training prepared by the researcher. In the training, the exercise will be demonstrated through demonstration method. Following training, women will be asked to perform progressive relaxation exercise at least 3 times a week (every other day). Women will be followed for 8 weeks with a progressive muscle relaxation exercise daily follow-up chart prepared by the researcher, and weekly reminders will be made (via WhatsApp® or text message). The final test will be administered to women online at the end of 8 weeks. RLS Severity Rating Scale form, Johns Hopkins Restless Legs Syndrome Quality of Life Scale and Pittsburg Sleep Quality Index will be used in the pre-test and post-test applications.
  Interventions: Behavioral: progressive muscle relaxation exercises
- no intervention (No Intervention): No intervention will be applied to women. Posttest application to women; It will be conducted online 8 weeks after the pre-test application. RLS Severity Rating Scale form, Johns Hopkins Restless Legs Syndrome Quality of Life Scale and Pittsburg Sleep Quality Index will be used in the pre-test and post-test applications.

INTERVENTIONS:
Behavioral: progressive muscle relaxation exercises — Progressive muscle relaxation exercises (PKGE); 16 large muscles (right hand and forearm, right upper arm, left hand and forearm of left arm, left upper arm, forehead, upper cheek and nose, chin, neck, abdomen, upper right arm, which people can do on their own after learning) leg, right calf, right foot, left upper leg, left thigh and left foot), followed by the contraction and then relaxation and accompanied by deep breathing, is a preferred method for reducing pain, anxiety and depression in individuals.The relaxation will be required to take 10-20 before stretching the next muscle group. In this way, the muscle groups in the hands, arms, neck, shoulder, chest, abdomen, hips, feet and fingers, face and the whole body will be voluntarily stretched and relaxed, and pregnant women will be relieved.
  Arms: progressive muscle relaxation exercises

SUMMARY:
Restless legs syndrome is a symptom that can be seen in all stages of a woman's life, but its frequency and severity increases with menopause. Restless legs syndrome is a neurological problem that occurs usually at night with an irresistible urge to move the legs. It is a progressive muscle relaxation exercise. Progressive muscle relaxation exercise is a systematic practice aimed at providing deep relaxation by exercising large muscle groups in the body along with breathing techniques. This study aims to evaluate the effect of progressive muscle relaxation exercise on the severity of restless legs syndrome, quality of life and sleep quality related to restless legs syndrome in menopausal women with restless legs syndrome.

DETAILED DESCRIPTION:
Menopause, which is a natural part of women's life; It is a condition that occurs between the ages of 45-52 on average and is characterized by hormonal changes and cessation of the menstrual cycle. Many symptoms are observed during menopause, such as hot flashes, sleep problems, mood disorders, sexual dysfunction, weight gain, and decline in cognitive functioning. Restless legs syndrome is another symptom that can be seen in all periods of a woman's life, but its frequency and severity increases with menopause. Restless legs syndrome is a neurological problem that occurs usually at night with an irresistible urge to move the legs. There are studies reporting that sleep problems, which are a common problem during the menopausal period, worsen with the addition of restless legs syndrome. Restless legs syndrome and sleep problems are two important factors that negatively affect the quality of life of women in the menopausal period. Alternative and complementary therapies are frequently used among the methods used to cope with menopausal symptoms and symptoms triggered by menopause. These methods include hypnosis, body-mind techniques, cognitive behavioral therapies, aromatherapies, and herbal supplements. It is stated that these techniques reduce the stress of women in the menopausal period and are effective in improving their quality of life. One of these methods is progressive muscle relaxation exercise. Progressive muscle relaxation exercise is a systematic practice that aims to provide deep relaxation by exercising large muscle groups in the body along with breathing techniques. There are studies reporting that PCGE is used effectively in coping with menopausal symptoms. This study aims to evaluate the effect of progressive muscle relaxation exercise on the severity of restless legs syndrome, quality of life and sleep quality related to restless legs syndrome in menopausal women with restless legs syndrome.

ELIGIBILITY:
Inclusion Criteria:

Having entered natural menopause

* At least 1 year has passed since the last menstrual period
* Not having any psychiatric disease
* Not having any communication problems (mental, auditory, visual, etc.)

Exclusion Criteria:

* Women not performing post-test applications
* Not doing progressive muscle relaxation exercises twice in a row.
* Wants to quit the research.
* The woman is hospitalized
* Inability to reach women during follow-ups

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Restless Legs Syndrome Severity | Change from Baseline RLS Severity at 8 weeks
  Measurements will be made using the RLS Severity Rating Scale. A total score is obtained, with the entire score range varying between 0 and 40; A score between 1-10 indicates mild disease, a score between 11-20 indicates moderate disease, a score between 21-30 indicates severe disease, and a score between 31-40 indicates very severe disease.
Quality of life associated with restless legs syndrome | Change from Baseline Quality of Life at 8 weeks
  Measurements will be made using the Johns Hopkins Restless Leg Syndrome Quality of Life Scale. The lowest score from the scale is 0 and the highest score is 100. As the score obtained from the scale decreases, it indicates that the quality of life associated with restless legs syndrome is poor.
Quality of sleep associated with restless legs syndrome | Change from Baseline Quality of Life at 8 weeks
  Measurements will be made using the Pittsburg Sleep Quality Index.A high total score indicates poor sleep quality. Total score is between 0-21. The index does not indicate the presence or frequency of sleep disturbances. However, a PSQI total score of 5 or above indicates poor sleep quality. The cut-off score indicating poor sleep quality is accepted as 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabük Training and Research Hospital, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR